CLINICAL TRIAL: NCT00560417
Title: A Randomized Trial Comparing Insulin Lispro Protamine Suspension With Insulin Glargine in Subjects With Type 2 Diabetes on Oral Antihyperglycemic Medications and Exenatide
Brief Title: Comparison of Two Basal Insulins for Patients With Type 2 Diabetes Taking Oral Diabetes Medicines and Exenatide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11647; F3Z-US-IOPB (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILPS (Active Comparator): Insulin Lispro Protamine Suspension (ILPS)
  Interventions: Drug: Insulin Lispro Protamine Suspension
- Glargine (Active Comparator): Insulin Glargine
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Lispro Protamine Suspension — Administered subcutaneously once a day at bedtime
  Other Names: LY275585[P]
  Arms: ILPS
Drug: Insulin Glargine — Administered subcutaneously once a day at bedtime
  Other Names: Lantus
  Arms: Glargine

SUMMARY:
This study will compare insulin lispro protamine suspension (ILPS) and insulin glargine in combination with the patient's oral diabetes medications and exenatide, for their ability to control blood sugar in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Must have type 2 diabetes
* Must be at least 18 years of age and less than 75 years of age
* Must be taking exenatide 10 micrograms twice a day (BID) for at least 3 months
* Must be taking one of the following oral diabetes medication regimens for at least 3 months: (1) metformin (2) metformin + sulfonylurea (3) metformin + thiazolidinedione (TZD). Doses must be at or above the following: Metformin--1500 mg/day, Sulfonylurea--1/2 the maximum daily dose according to the product label, TZD--30 mg/day pioglitazone
* Must have a hemoglobin A1C greater than or equal to 7.0% and less than or equal to 10.0%

Exclusion Criteria:

* Must not have used insulin on a regular basis during the past 2 years
* Must not have taken any glucose-lowering medications not included in the inclusion criteria in the past 3 months
* Must not have had more than one episode of severe hypoglycemia in the past 6 months
* Must not have clinically significant hematologic, oncologic, renal, cardiac, hepatic, or gastrointestinal disease
* Must not be pregnant or intend to get pregnant during the course of the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (49):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modesto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inverness, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Worth, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avon, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biddeford, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jefferson City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mason, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingsport, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Virginia Beach, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toa Baja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yabucoa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intention to Treat (ITT) Population consisted of all randomized participants who received at least one dose of study drug and had at least one post-baseline measurement.
Groups:
- ILPS: Insulin Lispro Protamine Suspension (ILPS) administered subcutaneously once a day at bedtime for 24 weeks
- Glargine: Insulin Glargine administered subcutaneously once a day at bedtime for 24 weeks
Period: Overall Study
Arm/Group | ILPS | Glargine
Started | 171 | 168
Intention to Treat (ITT) Population | 170 | 167
Completed | 154 | 151
Not Completed | 17 | 17
Not completed — Adverse Event | 3 | 2
Not completed — Entry Criteria Not Met | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 6
Not completed — Protocol Violation | 6 | 5
Not completed — Sponsor Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ILPS | Glargine | Total
Number analyzed (Participants) | 171 | 168 | 339
Age Continuous [Mean (Standard Deviation); unit: years] | 56.51 (9.73) | 56.24 (9.33) | 56.38 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 75 | 170
  Male | 76 | 93 | 169
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 13 | 14 | 27
  East Asian | 5 | 6 | 11
  Hispanic | 21 | 17 | 38
  Native American | 0 | 1 | 1
  West Asian (Indian sub-continent) | 2 | 0 | 2
  White | 130 | 130 | 260
Region of Enrollment [Number; unit: participants]
  United States | 165 | 165 | 330
  Puerto Rico | 6 | 3 | 9
Body Mass Index [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 34.92 (5.21) | 34.78 (5.17) | 34.85 (5.18)
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 101.57 (18.67) | 102.33 (19.73) | 101.95 (19.18)
Hemoglobin A1C [Mean (Standard Deviation); unit: percent of glycosylated hemoglobin] | 8.21 (0.79) | 8.22 (0.80) | 8.22 (0.79)
Sulfonylurea Group [Number; unit: participants] — Participants taking a sulfonylurea at baseline.
  participants
    Yes | 108 | 110 | 218
    No | 63 | 58 | 121
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.51 (5.98) | 10.31 (6.63) | 9.91 (6.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (HbA1c) at Endpoint (Last Observation Carried Forward [LOCF])
Description: Least squares mean values were controlled for Baseline + Baseline HbA1c Group + Baseline sulfonylurea (SU) Group.
Time Frame: Baseline, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: percent of glycosylated hemoglobin
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
percent of glycosylated hemoglobin
  Baseline | 8.48 (0.04) | 8.47 (0.04)
  Endpoint (LOCF) Change | -1.21 (0.07) | -1.43 (0.07)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Non-Inferiority or Equivalence — Noninferiority margin was prespecified at 0.4%; ANCOVA; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.06 to 0.38]

2. Secondary Outcome: Actual Hemoglobin A1C at 24 Weeks and Endpoint (LOCF)
Description: Least squares mean values were controlled for Baseline + Baseline HbA1c Group + Baseline SU Group.
Time Frame: 24 weeks, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: percent of glycosylated hemoglobin
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
percent of glycosylated hemoglobin
  24 weeks | 6.94 (0.07) | 6.70 (0.06)
  Endpoint (LOCF) | 7.00 (0.07) | 6.78 (0.07)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.003, ANCOVA — p-value is for 24 weeks; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.08 to 0.39]
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.008, ANCOVA — p-value is for Endpoint (LOCF); Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.06 to 0.38]

3. Secondary Outcome: Change From Baseline in Hemoglobin A1C at 24 Weeks and Endpoint (LOCF)
Description: Least squares mean values were controlled for Baseline + Baseline HbA1c Group + Baseline SU Group.
Time Frame: Baseline, 24 Weeks, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: percent of glycosylated hemoglobin
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
percent of glycosylated hemoglobin
  Baseline | 8.48 (0.04) | 8.47 (0.04)
  24 Weeks Change | -1.25 (0.07) | -1.49 (0.06)
  Endpoint (LOCF) Change | -1.21 (0.07) | -1.43 (0.07)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.003, ANCOVA — p-value is for 24 Weeks change; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.08 to 0.39]
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.008, ANCOVA — p-value is for Endpoint (LOCF) Change; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.06 to 0.38]

4. Secondary Outcome: Percentage of Participants With Hemoglobin A1C Less Than 7.0% and Hemoglobin A1C Less Than or Equal to 6.5%
Time Frame: Weeks 12, 18, 24 and Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Number; unit: percent of participants
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
percent of participants
  Week 12: HbA1c <7.0% | 46.9 | 50.7
  Week 12: HbA1c <=6.5% | 24.8 | 28.7
  Week 18: HbA1c <7.0% | 54.8 | 69.1
  Week 18: HbA1c <=6.5% | 30.8 | 37.6
  Week 24: HbA1c <7.0% | 55.4 | 63.4
  Week 24: HbA1c <=6.5% | 29.7 | 39.9
  Endpoint (LOCF): HbA1c <7.0% | 53.7 | 61.7
  Endpoint (LOCF): HbA1c <=6.5% | 28.4 | 38.9
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.561, Fisher Exact — p-value is for Week 12: HbA1c <7.0%
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.511, Fisher Exact — p-value is for Week 12: HbA1c <=6.5%
Statistical Analysis 3: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.012, Fisher Exact — p-value is for Week 18: HbA1c <7.0%
Statistical Analysis 4: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.269, Fisher Exact — p-value is for Week 18: HbA1c <=6.5%
Statistical Analysis 5: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.161, Fisher Exact — p-value is for Week 24: HbA1c <7.0%
Statistical Analysis 6: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.071, Fisher Exact — p-value is for Week 24: HbA1c <=6.5%
Statistical Analysis 7: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.177, Fisher Exact — p-value is for Endpoint (LOCF): HbA1c <7.0%
Statistical Analysis 8: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.060, Fisher Exact — p-value is for Endpoint (LOCF): HbA1c <=6.5%

5. Secondary Outcome: 7-Point Self-Monitored Blood Glucose (SMBG) Profiles at Baseline and Endpoint (LOCF)
Description: SMBG at morning pre-meal, morning post-prandial, midday pre-meal, midday post-prandial, evening pre-meal, evening postprandial, 0300 hours. Post-prandial glucose is measured 2 hours after the start of the meal.
Time Frame: Baseline, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
milligrams per deciliter (mg/dL)
  Baseline Morning Pre-Meal | 175.41 (39.54) | 180.86 (38.95)
  Baseline Morning Postprandial | 195.31 (54.65) | 190.84 (54.95)
  Baseline Midday Pre-Meal | 165.18 (43.51) | 166.34 (47.64)
  Baseline Midday Postprandial | 193.22 (46.95) | 200.25 (54.64)
  Baseline Evening Pre-Meal | 173.33 (44.60) | 175.14 (43.35)
  Baseline Evening Postprandial | 189.00 (49.62) | 184.92 (49.42)
  Baseline 0300 Hours | 170.51 (43.44) | 172.00 (39.10)
  Baseline Daily Mean 7-Point Blood Glucose | 180.19 (36.95) | 180.72 (38.17)
  Baseline Daily Mean Pre-Meal | 170.60 (36.06) | 172.66 (38.60)
  Baseline Daily Mean Postprandial | 192.37 (41.48) | 191.27 (46.11)
  Endpoint Morning Pre-Meal | 129.63 (31.58) | 127.01 (29.08)
  Endpoint Morning Postprandial | 152.32 (44.81) | 137.39 (36.65)
  Endpoint Midday Pre-Meal | 132.84 (36.63) | 129.71 (34.34)
  Endpoint Midday Postprandial | 161.77 (42.46) | 155.26 (37.86)
  Endpoint Evening Pre-Meal | 146.03 (37.93) | 135.93 (33.79)
  Endpoint Evening Postprandial | 159.14 (45.35) | 144.25 (34.17)
  Endpoint 0300 Hours | 123.96 (35.45) | 127.53 (30.90)
  Endpoint Daily Mean 7-Point Blood Glucose | 143.06 (30.00) | 136.17 (25.65)
  Endpoint Daily Mean Pre-Meal | 135.51 (30.39) | 129.32 (26.54)
  Endpoint Daily Mean Postprandial | 158.10 (36.81) | 146.12 (30.37)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.179, ANCOVA — p-value is for Endpoint Morning Pre-Meal; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 4.28, 95% CI 2-sided [-1.97 to 10.53]
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Endpoint Morning Postprandial; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 13.96, 95% CI 2-sided [5.72 to 22.19]
Statistical Analysis 3: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.325, ANCOVA — p-value is for Endpoint Midday Pre-Meal; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 3.80, 95% CI 2-sided [-3.79 to 11.39]
Statistical Analysis 4: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.051, ANCOVA — p-value is for Endpoint Midday Postprandial; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 8.73, 95% CI 2-sided [-0.04 to 17.50]
Statistical Analysis 5: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.003, ANCOVA — p-value is for Endpoint Evening Pre-Meal; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 10.92, 95% CI 2-sided [3.66 to 18.19]
Statistical Analysis 6: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.002, ANCOVA — p-value is for Endpoint Evening Postprandial; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 14.19, 95% CI 2-sided [5.44 to 22.94]
Statistical Analysis 7: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.415, ANCOVA — p-value is for Endpoint 0300 Hours; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = -3.03, 95% CI 2-sided [-10.35 to 4.28]
Statistical Analysis 8: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.015, ANCOVA — p-value is for Endpoint Daily Mean 7-Point Blood Glucose; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 7.39, 95% CI 2-sided [1.46 to 13.32]
Statistical Analysis 9: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.021, ANCOVA — p-value is for Endpoint Daily Mean Pre-Meal; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 7.12, 95% CI 2-sided [1.10 to 13.14]
Statistical Analysis 10: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Endpoint Daily Mean Postprandial; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 11.97, 95% CI 2-sided [5.01 to 18.93]

6. Secondary Outcome: Glycemic Variability at Baseline and Endpoint (LOCF)
Description: Glycemic variability was defined as the standard deviation (SD) of a participant's intra-day 7-point, self-monitored, blood glucose. Mean SD was calculated based on the SD for each participant in the study.
Time Frame: Baseline, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
mg/dL
  Baseline | 41.15 (13.69) | 39.02 (13.52)
  Endpoint | 36.78 (16.02) | 30.96 (13.24)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.131, ANOVA — p-value is for Baseline; Variable = Treatment + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [-0.68 to 5.22]
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p < 0.001, ANOVA — p-value is for Endpoint; Variable = Treatment + Baseline HbA1c Group + Baseline SU Group; Mean Difference (Final Values) = 5.99, 95% CI 2-sided [2.82 to 9.16]

7. Secondary Outcome: Incidence of Self-reported Hypoglycemic Episodes (All, Non-Nocturnal, Nocturnal, and Severe)
Description: Overall:any time after randomization.Episode:any time patient experienced sign/symptom associated with hypoglycemia, or had blood glucose level ≤70 mg/dL. Non-nocturnal:any episode that occurred between waking and bedtime. Nocturnal:any episode that occurred between bedtime and waking.Severe:episode with symptoms consistent with neuroglycopenia in which patient requires assistance,and is associated with:blood glucose value <50 mg/dL or prompt recovery after oral carbohydrate, glucagon, or intravenous glucose.Incidence(%)=(Number of patients experiencing episodes/number of patients in arm)*100.
Time Frame: Baseline to Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
percentage of participants
  All Reported - Endpoint | 41.8 | 43.1
  All Reported - Overall | 70.6 | 74.9
  Non-Nocturnal - Endpoint | 30.6 | 40.1
  Non-Nocturnal - Overall | 62.4 | 70.7
  Nocturnal - Endpoint | 21.8 | 11.4
  Nocturnal - Overall | 47.6 | 37.1
  Severe - Endpoint | 0 | 0
  Severe - Overall | 1.8 | 0
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.826, Fisher Exact — p-value is for all reported hypoglycemic events at endpoint
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.394, Fisher Exact — p-value is for all reported hypoglycemic events overall
Statistical Analysis 3: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.070, Fisher Exact — p-value is for non-nocturnal hypoglycemic events at endpoint
Statistical Analysis 4: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.133, Fisher Exact — p-value is for non-nocturnal hypoglycemic events overall
Statistical Analysis 5: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.013, Fisher Exact — p-value is for nocturnal hypoglycemic events at endpoint
Statistical Analysis 6: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.061, Fisher Exact — p-value is for nocturnal hypoglycemic events overall
Statistical Analysis 7: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.248, Fisher Exact — p-value is for severe hypoglycemic events overall

8. Secondary Outcome: Rate of All, Non-Nocturnal, and Nocturnal Self-Reported Hypoglycemic Episodes (Adjusted for One Year)
Description: Rate of self-reported hypoglycemic episodes, all, non-nocturnal, and nocturnal, at Endpoint (LOCF) and overall. Rate is reported as episodes/participant/365 days. Episode = any time participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a blood glucose level of ≤70 mg/dL, even if it was not associated with signs, symptoms, or treatment. Overall=any time during the post-randomization visits within the study period. Nocturnal=Any episode that occurs between bedtime and waking. Non-Nocturnal=Any episode that occurs between waking and bedtime.
Time Frame: Baseline to Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: episodes/participant/365 days
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
episodes/participant/365 days
  All reported episodes rate - Endpoint | 14.51 (27.75) | 15.29 (29.73)
  All reported episodes rate - Overall | 16.27 (23.19) | 18.05 (24.59)
  Non-Nocturnal reported episodes rate - Endpoint | 10.40 (23.46) | 13.20 (28.01)
  Non-Nocturnal reported episodes rate - Overall | 11.36 (19.16) | 14.83 (21.00)
  Nocturnal reported episodes rate - Endpoint | 4.01 (9.73) | 1.73 (5.53)
  Nocturnal reported episodes rate - Overall | 4.88 (8.43) | 3.01 (7.21)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.628, Negative Binomial regression model — p-value is for All reported episodes rate - Endpoint; Total hypoglycemia count=Treatment+Baseline HbA1c Group+Baseline SU Group with log of patient's total number of days of exposure as an offset variable
Statistical Analysis 2: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.570, Negative Binomial regression model — p-value is for All reported episodes rate - Overall; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.116, Negative Binomial regression model — p-value is for Non-Nocturnal reported episodes rate - Endpoint; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.044, Negative Binomial regression model — p-value is for Non-Nocturnal reported episodes rate - Overall; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.006, Negative Binomial regression model — p-value is for Nocturnal reported episodes rate - Endpoint; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.004, Negative Binomial regression model — p-value is for Nocturnal reported episodes rate - Overall; [statistical method as in outcome 8, analysis 1]

9. Secondary Outcome: Actual Body Weight at Baseline and Endpoint (LOCF)
Time Frame: Baseline, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
kilograms
  Baseline | 101.57 (18.67) | 102.62 (19.58)
  Endpoint | 101.85 (18.91) | 103.28 (19.42)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.343, ANCOVA — p-value is for endpoint; Variable = Treatment + Baseline + Baseline HbA1c Group + Baseline SU Group (Type III sums of squares)

10. Secondary Outcome: Change From Baseline in Body Weight at Endpoint (LOCF)
Time Frame: Baseline, Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 170 | 167
kilograms | 0.27 (3.38) | 0.66 (3.93)
Statistical Analysis 1: Comparison: ILPS; Test type: Superiority or Other; p = 0.417, t-test, 2 sided — p-value is for the change in body weight at endpoint in the ILPS treatment group
Statistical Analysis 2: Comparison: Glargine; Test type: Superiority or Other; p = 0.041, t-test, 2 sided — p-value is for the change in body weight at endpoint in the glargine treatment group
Statistical Analysis 3: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p = 0.343, ANOVA — p-value is for change in body weight at endpoint between ILPS and glargine treatment groups; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.15 to 0.40]

11. Secondary Outcome: Total Daily Insulin Dose at Endpoint (LOCF)
Time Frame: Endpoint (LOCF) up to 24 weeks
Population: All randomized participants with at least one post-baseline measurement. Intention to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Units of Insulin
Arm/Group | ILPS | Glargine
Number analyzed (Participants) | 168 | 165
Units of Insulin | 31.11 (18.87) | 37.93 (18.46)
Statistical Analysis 1: Comparison: ILPS vs Glargine; Test type: Superiority or Other; p < 0.001, ANOVA; Variable = Treatment + Baseline HbA1c Group+ Baseline SU Group

ADVERSE EVENTS:
Description: Adverse events are reported for the Intention to Treat (ITT) population.
Arm/Group | ILPS | Glargine
Serious Adverse Events (participants affected / at risk) | 9/170 | 5/167
Other Adverse Events (participants affected / at risk) | 96/170 | 115/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILPS (N=170) | Glargine (N=167)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis bacterial (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILPS (N=170) | Glargine (N=167)
Abdominal discomfort (Gastrointestinal disorders) | 6 (9) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (17) | 12 (31)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (14)
Nausea (Gastrointestinal disorders) | 13 (37) | 10 (14)
Vomiting (Gastrointestinal disorders) | 6 (7) | 8 (11)
Pyrexia (General disorders) | 1 (1) | 5 (5)
Bronchitis (Infections and infestations) | 1 (3) | 5 (9)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 12 (15)
Influenza (Infections and infestations) | 4 (8) | 3 (4)
Nasopharyngitis (Infections and infestations) | 12 (18) | 9 (14)
Sinusitis (Infections and infestations) | 7 (17) | 9 (26)
Upper respiratory tract infection (Infections and infestations) | 11 (23) | 10 (24)
Urinary tract infection (Infections and infestations) | 5 (9) | 2 (3)
Joint sprain (Injury, poisoning and procedural complications) | 4 (27) | 2 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (19) | 7 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (8) | 4 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 4 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 5 (17)
Headache (Nervous system disorders) | 11 (44) | 15 (42)
Sinus headache (Nervous system disorders) | 4 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 5 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 9 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 7 (11)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days